CLINICAL TRIAL: NCT00031954
Title: A Phase II Study Of Paclitaxel, Carboplatin And Gemcitabine In Previously Untreated Patients With Epithelial Ovarian Carcinoma FIGO Stage IIB-IV
Brief Title: Combination Chemotherapy in Treating Patients With Ovarian Epithelial, Fallopian Tube, or Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AGO Study Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGO-OVAR 8; AGOSG-OVAR-8; EU-20146
Record Dates: First submitted 2002-03-08; First posted 2003-07-01 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage II ovarian epithelial cancer; stage I ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Carboplatin; Gemcitabine; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have stage IC, stage IIB, stage III, or stage IV ovarian epithelial, fallopian tube, or peritoneal cancer that has not been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the tolerability and toxicity of paclitaxel, carboplatin, and gemcitabine in patients with previously untreated stage IC-IV ovarian epithelial, fallopian tube, or peritoneal carcinoma.
* Determine the response rate of patients treated with this regimen.
* Determine the time to progression and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30 minutes on day 1 and gemcitabine IV over 30-60 minutes on days 1 and 8. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3 and 6 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IC-IV ovarian epithelial, fallopian tube, or peritoneal carcinoma

  * No tumors of low-malignant potential (borderline tumors)
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 70-100%

Life expectancy:

* At least 6 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal

Renal:

* Glomerular filtration rate at least 60 mL/min

Cardiovascular:

* No history of congestive heart failure (New York Heart Association class III or IV heart disease) even if medically controlled
* No myocardial infarction within the past 6 months
* No history of atrial or ventricular arrhythmias

Neurologic:

* No history of seizure disorder
* No history of CNS disorder
* No pre-existing motor or sensory neuropathy or symptoms grade 2 or greater

Other:

* No severe concurrent infection
* No prior hypersensitivity reaction to products containing Cremophor EL or compounds chemically related to carboplatin, paclitaxel, or gemcitabine
* No complete bowel obstruction
* No other concurrent severe medical problems that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy
* No concurrent WBC transfusions

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy except replacement therapy or steroid antiemetics

Radiotherapy:

* No prior radiotherapy
* No concurrent radiotherapy

Surgery:

* No more than 6 weeks since prior definitive surgery

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2001-08; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of tolerability and toxicity of the combination therapy with paclitaxel, carboplatin and gemcitabine (P-C-G) in first line treatment of ovarian cancer patients. Evaluation of Drop-out rate due to toxicity | Based on decision level
  The decision level is reached, when the lower exact 95% confidence limit of the observed proportion is higher than the upper exact 95% confidence limit of the historical proportion, which corresponds to a power of 0.5 applying a significance level of 0.05

CONTACTS AND LOCATIONS:
Overall Officials: Andreas du Bois, MD, PhD, Study Chair — Dr. Horst-Schmidt-Kliniken
Locations (18):
- Germany (18):
  - Universitaetsklinikum Charite, Berlin
  - Zentralkrankenhaus, Bremen
  - Medizinische Klinik I, Dresden
  - Evangelisches Krankenhaus, Düsseldorf
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Staedtisches Krankenhaus FFM-Hoechst, Frankfurt am Main
  - Universitaetsklinik Goettingen, Göttingen
  - Klinik Fuer Innere Medizin Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Frauenklinik der MHH, Hanover
  - Vincentius Krankenhaus, Karlsruhe
  - Christian-Albrechts University of Kiel, Kiel
  - Klinik der Otto-v.-Guericke-Universitat, Magdeburg
  - Klinikum Grosshadern, Munich (Muenchen)
  - Klinikum Rechts Der Isar/Technische Universitaet Muenchen, Munich (Muenchen)
  - Klinik und Poliklinik fuer Kinderheilkunde, Münster
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaet Ulm, Ulm
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden

REFERENCES:
- [Result] du Bois A, Belau A, Wagner U, Pfisterer J, Schmalfeldt B, Richter B, Staehle A, Jackisch C, Lueck HJ, Schroeder W, Burges A, Olbricht S, Elser G; Arbeitsgemeinschaft Gynaekologische Onkologie Ovarian Cancer Study Group (AGO-OVAR). A phase II study of paclitaxel, carboplatin, and gemcitabine in previously untreated patients with epithelial ovarian cancer FIGO stage IC-IV (AGO-OVAR protocol OVAR-8). Gynecol Oncol. 2005 Feb;96(2):444-51. doi: 10.1016/j.ygyno.2004.10.020. PMID 15661234